CLINICAL TRIAL: NCT03455829
Title: Phase 1b/2 Safety, Pharmacokinetic, and Efficacy Study of G1T38 in Combination With Osimertinib in Patients With EGFR Mutation-Positive Metastatic Non-Small Cell Lung Cancer (NSCLC)
Brief Title: G1T38, a CDK 4/6 Inhibitor, in Combination With Osimertinib in EGFR-Mutant Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: G1 Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: G1T38-03; 2017-004315-39 (EudraCT Number)
Record Dates: First submitted 2018-02-28; First posted 2018-03-07 (Actual); Results first posted 2023-05-01 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Lung Cancer; Non-small Cell Lung Cancer
Keywords: Lung Cancer; Non-small Cell Lung Cancer; CDK 4/6 Inhibitor; EGFR-Positive; EGFR Mutation- Positive; T790M; EGFR Mutant; lerociclib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: Cohort 1 G1T38 + Osimertinib (Experimental): Patients will receive a single oral dose of G1T38 on Cycle 1 Day -16 and on Cycle 1 Day -2. Patients will receive oral osimertinib 80 mg beginning Cycle 1 Days -14. Patients will begin G1T38 once-daily dosing on Cycle 1 Day 1 (in combination with osimertinib 80 mg).
  Interventions: Drug: G1T38; Drug: Osimertinib
- Part 1: Cohort 2 G1T38 + Osimertinib (Experimental): Patients will receive a single oral dose of G1T38 on Cycle 1 Day -16 and on Cycle 1 Day -2. Patients will receive oral osimertinib 80 mg beginning Cycle 1 Days -14. Patients will begin G1T38 once-daily dosing on Cycle 1 Day 1 (in combination with osimertinib 80 mg).
  Interventions: Drug: G1T38; Drug: Osimertinib
- Part 1: Cohort 3 G1T38 + Osimertinib (Experimental): Patients will receive a single oral dose of G1T38 on Cycle 1 Day -16 and on Cycle 1 Day -2. Patients will receive oral osimertinib 80 mg beginning Cycle 1 Days -14. Patients will begin G1T38 once-daily dosing on Cycle 1 Day 1 (in combination with osimertinib 80 mg).
  Interventions: Drug: G1T38; Drug: Osimertinib
- Part 1: Cohort 4 G1T38 + Osimertinib (Experimental): Patients will receive a single oral dose of G1T38 on Cycle 1 Day -16 and on Cycle 1 Day -2. Patients will receive oral osimertinib 80 mg beginning Cycle 1 Days -14. Patients will begin G1T38 once-daily dosing on Cycle 1 Day 1 (in combination with osimertinib 80 mg).
  Interventions: Drug: G1T38; Drug: Osimertinib
- Part 1: Cohort 5 G1T38 + Osimertinib (Experimental): Patients will receive a single oral dose of G1T38 on Cycle 1 Day -16 and on Cycle 1 Day -2. Patients will receive oral osimertinib 80 mg beginning Cycle 1 Days -14. Patients will begin G1T38 once-daily dosing on Cycle 1 Day 1 (in combination with osimertinib 80 mg).
  Interventions: Drug: G1T38; Drug: Osimertinib

INTERVENTIONS:
Drug: G1T38 — CDK 4/6 inhibitor
  Other Names: Lerociclib
Drug: Osimertinib — EGFR TKI; 80 mg
  Other Names: Tagrisso

SUMMARY:
This was a study to investigate the potential clinical benefit of G1T38 as an oral therapy in combination with osimertinib in patients with EGFR mutation-positive metastatic non-small cell lung cancer.

The study was an open-label design, planned to consist of 2 parts: a safety, pharmacokinetic, and dose-finding portion (Part 1), and a randomized portion (Part 2). Both parts were to include 3 study phases: Screening Phase, Treatment Phase, and Survival Follow-up Phase. The Treatment Phase began on the day of first dose with study treatment and completes at the Post-Treatment Visit. Approximately, 144 patients were planned to be enrolled in the study.

DETAILED DESCRIPTION:
Part 2, the Phase 2 part of the study, was not conducted due to changes in corporate strategy. There were no safety signals identified in Phase 1/Part 1 that would have precluded the conduct of Part 2. As a result, 30 out of the planned 144 patients were enrolled.

All tumor assessments were conducted by the Investigators or site radiologist. In order to reduce the burden to the patients, data of overall survival (OS) were no longer required (since 29 January 2020). No OS analysis was conducted for Part 1 due to limited data in Part 1.

PK data for Cohorts 4 (150 BID) and 5 (200 BID) were not analyzed as they were deemed unnecessary, as the PK data from Cohorts 1-3 were sufficient to achieve the secondary study objective of assessing the effect of osimertinib on PK parameters of G1T38.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed EGFR mutation for non-small cell lung cancer associated with EGFR TKI sensitivity
* For Part 2, EGFR T790M mutation-positive tumor status
* Left ventricular ejection fraction (LVEF) ≥ institution's lower limit of the reference range
* For Part 1, evaluable or measurable disease as defined by RECIST, Version 1.1
* For Part 2, measurable disease as defined by RECIST, Version 1.1
* ECOG performance status 0 to 1
* Adequate organ function

Exclusion Criteria:

* Prior treatment with EGFR TKI within 9 days of first study dose
* For Part 1, prior treatment with more than 2 prior lines of chemotherapy for advanced NSCLC
* For Part 2, prior treatment with osimertinib or other T790M active EGFR TKI
* For Part 2, prior chemotherapy for advanced NSCLC
* Active uncontrolled/symptomatic CNS metastases, carcinomatous meningitis, or leptomeningeal disease
* Investigational drug within 3 months or 5 half-lives, whichever is longer, of first study dose
* Concurrent radiotherapy, radiotherapy within 28 days of first study dose, previous radiotherapy to the target lesion sites, or prior radiotherapy to > 25% of bone marrow
* Prior hematopoietic stem cell or bone marrow transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-29 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2022-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Contact, Study Director — G1 Therapeutics, Inc.
Locations (8):
- United States (8):
  - Beverly Hills Cancer Center, Beverly Hills, California
  - UCLA Medical Center, Division of Hematology/Oncology/Clinical Research Unit, Santa Monica, California
  - St Joseph Heritage Healthcare, Santa Rosa, California
  - Sylvester Comprehensive Cancer Center/University of Miami Miller School of Medicine Fox Building, Suite 200 G, Miami, Florida
  - Mofitt Cancer Center, Tampa, Florida
  - Univ. of Michigan Hospitals, Ann Arbor, Michigan
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: Cohort 1 Lerociclib at 200 mg QD: Part 1: G1T38/Lerociclib at 200 mg once daily (QD) orally + Osimertinib 80 mg once daily (QD) orally
- Part 1: Cohort 2 Lerociclib at 300 mg QD: Part 1: G1T38/Lerociclib at 300 mg once daily (QD) orally + Osimertinib 80 mg once daily (QD) orally
- Part 1: Cohort 3 Lerociclib at 400 mg QD: Part 1: G1T38/Lerociclib at 400 mg once daily (QD) orally + Osimertinib 80 mg once daily (QD) orally
- Part 1: Cohort 4 Lerociclib at 150 mg BID: Part 1: G1T38/Lerociclib at 150 mg twice daily (BID) orally + Osimertinib 80 mg once daily (QD) orally
- Part 1: Cohort 5 Lerociclib at 200 mg BID: Part 1: G1T38/Lerociclib at 200 mg twice daily (BID) orally + Osimertinib 80 mg once daily (QD) orally
Period: Overall Study
Arm/Group | Part 1: Cohort 1 Lerociclib at 200 mg QD | Part 1: Cohort 2 Lerociclib at 300 mg QD | Part 1: Cohort 3 Lerociclib at 400 mg QD | Part 1: Cohort 4 Lerociclib at 150 mg BID | Part 1: Cohort 5 Lerociclib at 200 mg BID
Started | 7 | 6 | 4 | 7 | 6
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 6 | 4 | 7 | 6
Not completed — Death | 2 | 3 | 2 | 4 | 2
Not completed — Study terminated and patients did not have progressive disease or died | 5 | 3 | 2 | 2 | 3
Not completed — Disease progression | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All enrolled patients who were administered at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Cohort 1 Lerociclib at 200 mg QD | Part 1: Cohort 2 Lerociclib at 300 mg QD | Part 1: Cohort 3 Lerociclib at 400 mg QD | Part 1: Cohort 4 Lerociclib at 150 mg BID | Part 1: Cohort 5 Lerociclib at 200 mg BID | Total
Number analyzed (Participants) | 7 | 6 | 4 | 7 | 6 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.71 (11.265) | 62.67 (8.779) | 62.75 (7.805) | 61.43 (15.757) | 66.17 (3.764) | 63.10 (10.118)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 3 | 5 | 4 | 21
  Male | 1 | 3 | 1 | 2 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 0 | 1 | 0 | 4
  Not Hispanic or Latino | 3 | 6 | 3 | 5 | 6 | 23
  Unknown or Not Reported | 1 | 0 | 1 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 1 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 2 | 1 | 3
  White | 1 | 5 | 2 | 3 | 4 | 15
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 0 | 1 | 2 | 0 | 8

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity
Description: The percentage of patients experiencing DLTs in Part 1 of the study in each cohort, including:
  * Grade 4 neutropenia
  * ≥ Grade 3 neutropenic infection/febrile neutropenia
  * Grade 4 thrombocytopenia
  * ≥ Grade 3 thrombocytopenia with bleeding
  * ≥ Grade 3 nonhematologic toxicity (additional criteria for nausea, vomiting, diarrhea, or fatigue: lasting > 5 days with maximal medical management)
  * Liver function test abnormalities meeting Hy's Law criteria (aspartate aminotransferase [AST] or alanine aminotransferase [ALT] ≥ 3 × upper limit of normal [ULN] and total bilirubin ≥ 2 × ULN).
Time Frame: Cycle 1 Day -16 to Cycle 1 Day 28
Population: Safety analysis set: including all enrolled patients who were administered at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1 Lerociclib at 200 mg QD | Part 1: Cohort 2 Lerociclib at 300 mg QD | Part 1: Cohort 3 Lerociclib at 400 mg QD | Part 1: Cohort 4 Lerociclib at 150 mg BID | Part 1: Cohort 5 Lerociclib at 200 mg BID
Number analyzed (Participants) | 7 | 6 | 4 | 7 | 6
Participants | 0 | 0 | 1 | 0 | 0

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Median time (months) and 95% CI from date of first dose of study drug/randomization until date of documented disease progression or death due to any cause.
  Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1 guidelines for tumor assessments were used to determine progression. Progressive Disease (PD) was defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: 36 months
Population: Full Analysis Set: All enrolled patients who were administered at least one dose of continuous daily G1T38.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: Cohort 1 Lerociclib at 200 mg QD | Part 1: Cohort 2 Lerociclib at 300 mg QD | Part 1: Cohort 3 Lerociclib at 400 mg QD | Part 1: Cohort 4 Lerociclib at 150 mg BID | Part 1: Cohort 5 Lerociclib at 200 mg BID
Number analyzed (Participants) | 7 | 6 | 4 | 6 | 6
months | 19.3 [2.0 to NA] — The upper confidence limit for the median was not estimable, as the upper confidence limits for the survivor function lies above 0.5. | 6.0 [1.8 to NA] — The upper confidence limit for the median was not estimable, as the upper confidence limits for the survivor function lies above 0.5. | 1.4 [0.7 to NA] — The upper confidence limit for the median was not estimable, as the upper confidence limits for the survivor function lies above 0.5. | 7.2 [1.6 to NA] — The upper confidence limit for the median was not estimable, as the upper confidence limits for the survivor function lies above 0.5. | 12.9 [3.6 to NA] — The upper confidence limit for the median was not estimable, as the upper confidence limits for the survivor function lies above 0.5.

3. Secondary Outcome: Best Overall Tumor Response
Description: The percentage of patients who fall into each category of Best overall response (BOR) as defined by Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1 guidelines.
  Complete Response (CR): Disappearance of all target lesions. Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions.
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
  When no imaging/measurement is done, the patient is not evaluable (NE); and if only a subset of lesion measurements are made, usually the case is also considered NE.
Time Frame: 21 months
Population: The response evaluable analysis set includes all patients who received study drug, had a measurable lesion (target lesions) at the baseline tumor assessment, and either (i) had at least 1 post-baseline tumor assessment, or (ii) did not have a post-baseline tumor assessment but had clinical progression as noted by the investigator, or died due to disease progression before their first post-baseline tumor scan.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Cohort 1 Lerociclib at 200 mg QD | Part 1: Cohort 2 Lerociclib at 300 mg QD | Part 1: Cohort 3 Lerociclib at 400 mg QD | Part 1: Cohort 4 Lerociclib at 150 mg BID | Part 1: Cohort 5 Lerociclib at 200 mg BID
Number analyzed (Participants) | 6 | 6 | 4 | 7 | 5
Participants
  Complete Response (CR) | 0 | 0 | 0 | 0 | 0
  Partial Response (PR) | 2 | 1 | 0 | 1 | 3
  Stable Disease (SD) | 2 | 4 | 1 | 3 | 0
  Progressive Disease (PD) | 1 | 1 | 3 | 2 | 1
  Not Evaluable (NE) | 1 | 0 | 0 | 1 | 1

4. Secondary Outcome: Pharmacokinetics of G1T38 and Metabolite G1T30: Maximum Plasma Concentration (Cmax)
Description: The observed peak plasma concentration determined from the plasma concentration versus time data.
Time Frame: Part 1, Cycle 1 Day -16 to Day -2.
Population: The analysis population included only those patients that received G1T38 on a once daily schedule, that is Cohorts 1-3. Pharmacokinetic data for Cohorts 4 and 5 were not collected due to the twice daily dosing schedule implemented, per recommendation of the Safety Monitoring Committee, for these 2 cohorts.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Part 1: Cohort 1 Lerociclib at 200 mg QD | Part 1: Cohort 2 Lerociclib at 300 mg QD | Part 1: Cohort 3 Lerociclib at 400 mg QD
Number analyzed (Participants) | 7 | 4 | 4
ng/mL
  G1T38 Cycle 1 Day -16 | 27.229 (8.936) | 33.375 (12.212) | 43.850 (21.942)
  G1T38 Cycle 1 Day -2 | 17.257 (1.471) | 26.400 (2.689) | 42.700 (25.107)
  Metabolite G1T30 Cycle 1 Day -16 | 3.080 (1.301) | 3.568 (0.633) | 4.220 (1.717)
  Metabolite G1T30 Cycle 1 Day -2 | 2.736 (0.764) | 3.853 (1.146) | 5.970 (4.369)

5. Secondary Outcome: Pharmacokinetics of G1T38 and Metabolite G1T30: Area Under Curve - Plasma Concentration (AUC) Infinity
Description: Area under the concentration-time curve from time zero extrapolated to infinity using the linear-up log-down trapezoidal rule.
Time Frame: Part 1, Cycle 1 Day -16 to Day -2.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Part 1: Cohort 1 Lerociclib at 200 mg QD | Part 1: Cohort 2 Lerociclib at 300 mg QD | Part 1: Cohort 3 Lerociclib at 400 mg QD
Number analyzed (Participants) | 7 | 4 | 4
h*ng/mL
  G1T38 Cycle 1 Day -16 | 319.6 (107) | 391.0 (85.6) | 715.6 (359)
  G1T38 Cycle 1 Day -2 | 277.4 (63.2) | 390.0 (91.0) | 802.3 (519)
  Metabolite G1T30 Cycle 1 Day -16 | 28.443 (17.175) | 30.853 (10.577) | 53.971 (23.638)
  Metabolite G1T30 Cycle 1 Day -2 | 30.110 (11.255) | 44.745 (13.929) | 80.145 (66.239)

6. Secondary Outcome: Pharmacokinetics of G1T38 and Metabolite G1T30: Plasma: Terminal Half Life (T1/2)
Description: Terminal half-life, defined as 0.693 divided by the terminal phase rate constant by λz , determined by linear regression of at least 3 points on the terminal phase of the log-linear plasma concentration-time curve.
Time Frame: Part 1, Cycle 1 Day -16 to Day -2.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Part 1: Cohort 1 Lerociclib at 200 mg QD | Part 1: Cohort 2 Lerociclib at 300 mg QD | Part 1: Cohort 3 Lerociclib at 400 mg QD
Number analyzed (Participants) | 7 | 4 | 4
hour
  G1T38 Cycle 1 Day -16 | 13.83 (1.95) | 16.30 (4.36) | 15.59 (2.12)
  G1T38 Cycle 1 Day -2 | 13.59 (2.88) | 12.61 (1.71) | 13.93 (2.14)
  Metabolite G1T30 Cycle 1 Day -16 | 11.771 (7.248) | 12.238 (8.072) | 22.614 (3.297)
  Metabolite G1T30 Cycle 1 Day -2 | 13.722 (8.025) | 18.220 (2.027) | 18.582 (2.977)

7. Secondary Outcome: Pharmacokinetics of G1T38: Plasma - Volume of Distribution
Description: Volume of distribution in the terminal elimination phase, calculated as:
  Vz/F = (CL/F)/λz
Time Frame: Part 1, Cycle 1 Day -16 to Day -2.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Liter
Arm/Group | Part 1: Cohort 1 Lerociclib at 200 mg QD | Part 1: Cohort 2 Lerociclib at 300 mg QD | Part 1: Cohort 3 Lerociclib at 400 mg QD
Number analyzed (Participants) | 7 | 4 | 4
Liter
  G1T38 Cycle 1 Day -16 | 14000 (6540) | 18700 (6910) | 15900 (9210)
  G1T38 Cycle 1 Day -2 | 14900 (4660) | 14800 (5060) | 12900 (6490)

ADVERSE EVENTS:
Time Frame: The SAE reporting period started at the time of informed consent and the AE reporting period started from the time of first dose of study drug; both were assessed through 30 calendar days after the last administration of lerociclib/osimertnib, an average of 11 months for each participant (Mean exposure + 30 days/1 month).
Description: An AE is defined as any untoward medical occurrence in a patient administered a medicinal product that does not necessarily have a causal relationship with this treatment, but does not include Progression of the malignancy under study. Deaths which were unequivocally due to disease progression, were documented in the eCRF module, but were not reported as SAEs during the study.
Arm/Group | Part 1: Cohort 1 Lerociclib at 200 mg QD | Part 1: Cohort 2 Lerociclib at 300 mg QD | Part 1: Cohort 3 Lerociclib at 400 mg QD | Part 1: Cohort 4 Lerociclib at 150 mg BID | Part 1: Cohort 5 Lerociclib at 200 mg BID
All-Cause Mortality (participants affected / at risk) | 2/7 | 3/6 | 2/4 | 4/7 | 2/6
Serious Adverse Events (participants affected / at risk) | 2/7 | 1/6 | 1/4 | 0/7 | 2/6
Other Adverse Events (participants affected / at risk) | 7/7 | 6/6 | 4/4 | 7/7 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Cohort 1 Lerociclib at 200 mg QD (N=7) | Part 1: Cohort 2 Lerociclib at 300 mg QD (N=6) | Part 1: Cohort 3 Lerociclib at 400 mg QD (N=4) | Part 1: Cohort 4 Lerociclib at 150 mg BID (N=7) | Part 1: Cohort 5 Lerociclib at 200 mg BID (N=6)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Cohort 1 Lerociclib at 200 mg QD (N=7) | Part 1: Cohort 2 Lerociclib at 300 mg QD (N=6) | Part 1: Cohort 3 Lerociclib at 400 mg QD (N=4) | Part 1: Cohort 4 Lerociclib at 150 mg BID (N=7) | Part 1: Cohort 5 Lerociclib at 200 mg BID (N=6)
Anaemia (Blood and lymphatic system disorders) | 5 (34) | 2 (4) | 2 (3) | 1 (5) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 4 (35) | 2 (7) | 1 (1) | 1 (2) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (22) | 3 (7) | 1 (1) | 2 (4) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 3 (13) | 1 (4) | 1 (1) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 (3) | 3 (4) | 1 (3) | 1 (3) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 5 (18) | 6 (13) | 4 (10) | 6 (6) | 6 (11)
Nausea (Gastrointestinal disorders) | 5 (10) | 5 (7) | 3 (6) | 2 (2) | 3 (3)
Vomiting (Gastrointestinal disorders) | 5 (7) | 4 (5) | 2 (4) | 1 (1) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 3 (7) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (5) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 2 (3) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal incontinence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glossodynia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue coated (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 5 (15) | 1 (5) | 2 (16) | 2 (7) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (4) | 0 (0) | 1 (2) | 1 (1) | 1 (2)
Lymphocyte count decreased (Investigations) | 3 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 4 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 2 (4) | 1 (3) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Blood creatinine increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 4 (23) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (4) | 1 (1) | 0 (0) | 2 (3) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (5) | 1 (1) | 2 (2) | 2 (2) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 2 (3) | 0 (0) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 2 (6) | 1 (3) | 2 (4) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 3 (5) | 0 (0) | 3 (3) | 2 (2)
Chills (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0)
Secretion discharge (General disorders) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Early satiety (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 5 (6) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0) | 1 (2) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Altered state of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 3 (5) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Xeroderma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Glycosuria (Renal and urinary disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctival haemorrhage (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual impairment (Eye disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vitreous detachment (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Corneal abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic steatosis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
A limitation of the trial is small numbers of subjects, since only the Phase 1/Part 1 part of the trial was conducted.

A lack of a control group, blinding and randomization also limits the utility of the information, so it is difficult to determine if there is any change in safety or tolerability of the combination of G1T38 + osimertinib from that of osimertinib alone or if there was any selection bias introduced.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-09-02): https://cdn.clinicaltrials.gov/large-docs/29/NCT03455829/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT03455829/SAP_001.pdf